CLINICAL TRIAL: NCT02153398
Title: An Open-label, Parallel-group, Multi-centre, Phase I/III Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of Repeated Once-daily Oral Administration of D961H 10 mg and D961H 20 mg in Japanese Paediatric Patients 1 to 14 Years Old With Gastrointestinal Acid Related Diseases
Brief Title: A Phase I/III Study of D961H 10 mg and 20 mg in Japanese Paediatric Patients With Gastrointestinal Acid Related Diseases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D961TC00002; 26-022 (Other: PMDA)
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-11

CONDITIONS: Gastric Ulcer (GU); Duodenal Ulcer (DU); Anastomotic Ulcer (AU); Non-erosive Reflux Esophagitis Disease (NERD); Reflux Esophagitis (RE); Zollinger-Ellison Syndrome
Keywords: Gastric ulcer (GU); Duodenal ulcer (DU); Anastomotic ulcer (AU); Non-erosive reflux esophagitis disease (NERD); Reflux esophagitis (RE); Zollinger-Ellison syndrome
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer; Esophagitis, Peptic; Zollinger-Ellison Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1: D961H sachet 10 mg (Experimental): Age: ≥1 year Weight: <20 kg
  Interventions: Drug: D961H sachet 10 mg
- Group 2: D961H capsule 10mg (Experimental): Age: ≥1 year to 11years Weight: ≥20 kg
  Interventions: Drug: D961H capsule 10mg
- Group 3: D961H capsule 20 mg (Experimental): Age: ≥1 year to 11years Weight: ≥20 kg
  Interventions: Drug: D961H capsule 20 mg
- Group 4: D961H capsule 10 mg (Experimental): Age: 12 to 14 years Weight: ≥20 kg
  Interventions: Drug: D961H capsule 10mg
- Group 5: D961H capsule 20 mg (Experimental): Age: 12 to 14 years Weight: ≥20 kg
  Interventions: Drug: D961H capsule 20 mg

INTERVENTIONS:
Drug: D961H sachet 10 mg
  Arms: Group 1: D961H sachet 10 mg
Drug: D961H capsule 10mg
  Arms: Group 2: D961H capsule 10mg; Group 4: D961H capsule 10 mg
Drug: D961H capsule 20 mg
  Arms: Group 3: D961H capsule 20 mg; Group 5: D961H capsule 20 mg

SUMMARY:
The objective of this study is to assess the safety, pharmacokinetics, pharmacodynamics and efficacy of repeated once daily oral administration of D961H 10 mg and D961H 20 mg in Japanese paediatric patients aged 1 to 14 years old who either have a diagnosis of or are suspected to have gastric ulcer (GU), duodenal ulcer (DU), anastomotic ulcer (AU), non-erosive reflux esophagitis disease (NERD), reflux esophagitis (RE) or Zollinger-Ellison syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent from the patient's guardian
* Patients aged ≥ 1 year to 14 years old
* Patients who have a diagnosis of or suspected to have GU, DU, AU, NERD, RE or Zollinger-Ellison syndrome.

Exclusion Criteria:

* Patients less than 10 kg in weight.
* Use of any other investigational compounds or participations in another clinical trial within 4 weeks prior to the randomisation/registration.
* Significant clinical illness within 4 weeks prior to the registration
* Presence of hepatic diseases or other conditions that could interfere with evaluation of the study as judged by the investigators.
* Positive for pregnancy test by urinary or lactation for post-menarchal females.
* Previous total gastrectomy

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- Japan (15):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Izumi-shi
  - Research Site, Maebashi
  - Research Site, Matsumoto-shi
  - Research Site, Osaka
  - Research Site, Saitama-shi
  - Research Site, Sapporo
  - Research Site, Setagaya-ku
  - Research Site, Shimotsuke-shi
  - Research Site, Shinjuku-ku
  - Research Site, Suzaka-shi
  - Research Site, Ureshino-shi
  - Research Site, Yokohama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled on 24 June 2014 Last subject last visit on 04 April 2016. This study was conducted at a total of 20 sites in Japan.
Pre-assignment Details: Out of 55 enrolled subjects, 50 subjects were registered and 5 subjects were not registered. The reason of no registration was 'Did not meet inclusion/exclusion criteria' (5 subjects).
Groups:
- Group 1: D961H sachet 10 mg Age: 1-11 years and Weight: <20 kg
- Group 2: D961H capsule 10 mg Age: 1-11 years and Weight: ≥20 kg
- Group 3: D961H capsule 20 mg Age: 1-11 years and Weight: ≥20 kg
- Group 4: D961H capsule 10 mg Age: 12-14 years and Weight: ≥20 kg
- Group 5: D961H capsule 20 mg Age: 12-14 years and Weight: ≥20 kg
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Started | 10 | 10 | 10 | 10 | 10
Completed | 9 | 10 | 9 | 9 | 10
Not Completed | 1 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.6 (2.2) | 8.9 (0.7) | 8.4 (1.8) | 13.4 (0.7) | 13.1 (0.9) | 9.5 (3.9)
Age, Customized [Number; unit: Participants]
  <= 3 years | 5 | 0 | 0 | 0 | 0 | 5
  4-5 years | 2 | 0 | 0 | 0 | 0 | 2
  6-7 years | 3 | 0 | 4 | 0 | 0 | 7
  8-9 years | 0 | 8 | 3 | 0 | 0 | 11
  10-11 years | 0 | 2 | 3 | 0 | 0 | 5
  12-14 years | 0 | 0 | 0 | 10 | 10 | 20
Gender [Count of Participants; unit: Participants]
  Female | 5 | 6 | 2 | 7 | 6 | 26
  Male | 5 | 4 | 8 | 3 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Disappearance of Heartburn at Week 8 by Patient Diaries
Description: The disappearance of heartburn was assessed by the intensity of the symptom at Week 8. Patients who recognized disappearance of heartburn were defined as those who selected "Mild", "Moderate", or "Severe" to the question about the intensity in the patient diary at pre-dose and had the maximum intensity of "None" at Week 8.
Time Frame: 8 weeks
Population: Participants who had heartburn at pre-dose in patient diary and obtained available diary data at Week 8.
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 2 | 3 | 1 | 1 | 4
Participants | 2 | 0 | 0 | 1 | 3

2. Primary Outcome: Disappearance of Epigastric Pain at Week 8 by Patient Diaries
Description: The disappearance of epigastric pain was assessed by the intensity of the symptom at Week 8. Patients who recognized disappearance of epigastric pain were defined as those who selected "Mild", "Moderate", or "Severe" to the question about the intensity in the patient diary at pre-dose and had the maximum intensity of "None" at Week 8.
Time Frame: 8 weeks
Population: Participants who had epigastric pain at pre-dose in patient diary and obtained available diary data at Week 8.
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 2 | 6 | 5 | 4 | 7
Participants | 2 | 3 | 5 | 1 | 3

3. Primary Outcome: Disappearance of Upper Abdominal Discomfort at Week 8 by Patient Diaries
Description: The disappearance of upper abdominal discomfort was assessed by the intensity of the symptom at Week 8. Patients who recognized disappearance of upper abdominal discomfort were defined as those who selected "Mild", "Moderate", or "Severe" to the question about the intensity in the patient diary at pre-dose and had the maximum intensity of "None" at Week 8.
Time Frame: 8 weeks
Population: Participants who had upper abdominal discomfort at pre-dose in patient diary and obtained available diary data at Week 8.
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 3 | 6 | 4 | 4 | 6
Participants | 3 | 2 | 4 | 2 | 2

4. Primary Outcome: Disappearance of Regurgitation at Week 8 by Patient Diaries
Description: The disappearance of regurgitation was assessed by the intensity of the symptom at Week 8. Patients who recognized disappearance of regurgitation were defined as those who selected "Mild", "Moderate", or "Severe" to the question about the intensity in the patient diary at pre-dose and had the maximum intensity of "None" at Week 8.
Time Frame: 8 weeks
Population: Participants who had regurgitation at pre-dose in patient diary and obtained available diary data at Week 8.
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 4 | 3 | 5 | 3 | 4
Participants | 3 | 2 | 3 | 2 | 4

5. Primary Outcome: Aggravation of Heartburn at Week 8 by Patient Diaries
Description: The aggravation of heartburn was assessed by the intensity of the symptom at Week 8. Patients who recognized aggravation of heartburn were defined as those who selected "None" to the question about the intensity in the patient diary at pre-dose and had the maximum intensity of "Mild", "Moderate" or "Severe" at Week 8.
Time Frame: 8 weeks
Population: Participants who had no heartburn at pre-dose in patient diary and obtained available diary data at Week 8.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 7 | 7 | 8 | 8 | 6
participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Aggravation of Epigastric Pain at Week 8 by Patient Diaries
Description: The aggravation of epigastric pain was assessed by the intensity of the symptom at Week 8. Patients who recognized aggravation of epigastric pain were defined as those who selected "None" to the question about the intensity in the patient diary at pre-dose and had the maximum intensity of "Mild", "Moderate" or "Severe" at Week 8.
Time Frame: 8 weeks
Population: Participants who had no epigastric pain at pre-dose in patient diary and obtained available diary data at Week 8.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 7 | 4 | 4 | 5 | 3
participants | 0 | 0 | 1 | 1 | 1

7. Primary Outcome: Aggravation of Upper Abdominal Discomfort at Week 8 by Patient Diaries
Description: The aggravation of upper abdominal discomfort was assessed by the intensity of the symptom at Week 8. Patients who recognized aggravation of upper abdominal discomfort were defined as those who selected "None" to the question about the intensity in the patient diary at pre-dose and had the maximum intensity of "Mild", "Moderate" or "Severe" at Week 8.
Time Frame: 8 weeks
Population: Participants who had no upper abdominal discomfort at pre-dose in patient diary and obtained available diary data at Week 8.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 6 | 4 | 5 | 5 | 4
participants | 0 | 0 | 2 | 1 | 0

8. Primary Outcome: Aggravation of Regurgitation at Week 8 by Patient Diaries
Description: The aggravation of regurgitation was assessed by the intensity of the symptom at Week 8. Patients who recognized aggravation of regurgitation were defined as those who selected "None" to the question about the intensity in the patient diary at pre-dose and had the maximum intensity of "Mild", "Moderate" or "Severe" at Week 8.
Time Frame: 8 weeks
Population: Participants who had no regurgitation at pre-dose in patient diary and obtained available diary data at Week 8.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 5 | 7 | 4 | 6 | 6
participants | 2 | 0 | 1 | 0 | 0

9. Primary Outcome: Disappearance of Heartburn at Week 8 by Investigators
Description: The investigators assessed the presence/absence and the intensity of heartburn at baseline and Week 8 based on questioning the patients or patients' guardians and the patient diary. Patients who recognized disappearance of heartburn were defined as those who had a heartburn at pre-dose and did not have the corresponding symptoms at Week 8 judged by investigators.
Time Frame: 8 weeks
Population: Participants who had a heartburn at pre-dose and were evaluated the symptom at Week 8 by investigators.
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 2 | 2 | 0 | 2 | 3
Participants | 2 | 1 |  | 2 | 2

10. Primary Outcome: Disappearance of Epigastric Pain at Week 8 by Investigators
Description: The investigators assessed the presence/absence and the intensity of epigastric pain at baseline and Week 8 based on questioning the patients or patients' guardians and the patient diary. Patients who recognized disappearance of epigastric pain were defined as those who had an epigastric pain at pre-dose and did not have the corresponding symptoms at Week 8 judged by investigators.
Time Frame: 8 weeks
Population: Participants who had an epigastric pain at pre-dose and were evaluated the symptom at Week 8 by investigators.
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 2 | 6 | 4 | 7 | 9
Participants | 2 | 5 | 4 | 2 | 6

11. Primary Outcome: Disappearance of Upper Abdominal Discomfort at Week 8 by Investigators
Description: The investigators assessed the presence/absence and the intensity of upper abdominal discomfort at baseline and Week 8 based on questioning the patients or patients' guardians and the patient diary. Patients who recognized disappearance of upper abdominal discomfort were defined as those who had an upper abdominal discomfort at pre-dose and did not have the corresponding symptoms at Week 8 judged by investigators.
Time Frame: 8 weeks
Population: Participants who had an upper abdominal discomfort at pre-dose and were evaluated the symptom at Week 8 by investigators.
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 3 | 6 | 5 | 7 | 6
Participants | 3 | 5 | 4 | 4 | 3

12. Primary Outcome: Disappearance of Regurgitation at Week 8 by Investigators
Description: The investigators assessed the presence/absence and the intensity of regurgitation at baseline and Week 8 based on questioning the patients or patients' guardians and the patient diary. Patients who recognized disappearance of regurgitation were defined as those who had a regurgitation at pre-dose and did not have the corresponding symptoms at Week 8 judged by investigators.
Time Frame: 8 weeks
Population: Participants who had a regurgitation at pre-dose and were evaluated the symptom at Week 8 by investigators.
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 4 | 1 | 5 | 1 | 3
Participants | 3 | 0 | 3 | 1 | 3

13. Primary Outcome: Aggravation of Heartburn at Week 8 by Investigators
Description: The investigators assessed the presence/absence and the intensity of heartburn at baseline and Week 8 based on questioning the patients or patients' guardians and the patient diary. Patients who recognized aggravation of heartburn were defined as those who had no heartburn at pre-dose and did have any of the corresponding symptoms at Week 8 judged by investigators.
Time Frame: 8 weeks
Population: Participants who had no heartburn at pre-dose and were evaluated the symptom at Week 8 by investigators.
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 7 | 8 | 9 | 7 | 7
Participants | 0 | 0 | 0 | 1 | 0

14. Primary Outcome: Aggravation of Epigastric Pain at Week 8 by Investigators
Description: The investigators assessed the presence/absence and the intensity of epigastric pain at baseline and Week 8 based on questioning the patients or patients' guardians and the patient diary. Patients who recognized aggravation of epigastric pain were defined as those who had no epigastric pain at pre-dose and did have any of the corresponding symptoms at Week 8 judged by investigators.
Time Frame: 8 weeks
Population: Participants who had no epigastric pain at pre-dose and were evaluated the symptom at Week 8 by investigators.
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 7 | 4 | 5 | 2 | 1
Participants | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Aggravation of Upper Abdominal Discomfort at Week 8 by Investigators
Description: The investigators assessed the presence/absence and the intensity of upper abdominal discomfort at baseline and Week 8 based on questioning the patients or patients' guardians and the patient diary. Patients who recognized aggravation of upper abdominal discomfort were defined as those who had no upper abdominal discomfort at pre-dose and did have any of the corresponding symptoms at Week 8 judged by investigators.
Time Frame: 8 weeks
Population: Participants who had no upper abdominal discomfort at pre-dose and were evaluated the symptom at Week 8 by investigators.
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 6 | 4 | 4 | 2 | 4
Participants | 0 | 0 | 0 | 1 | 0

16. Primary Outcome: Aggravation of Regurgitation at Week 8 by Investigators
Description: The investigators assessed the presence/absence and the intensity of regurgitation at baseline and Week 8 based on questioning the patients or patients' guardians and the patient diary. Patients who recognized aggravation of regurgitation were defined as those who had no regurgitation at pre-dose and did have any of the corresponding symptoms at Week 8 judged by investigators.
Time Frame: 8 weeks
Population: Participants who had no regurgitation at pre-dose and were evaluated the symptom at Week 8 by investigators.
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 5 | 9 | 4 | 8 | 7
Participants | 0 | 0 | 1 | 0 | 1

17. Secondary Outcome: Area Under the Plasma Concentration-time Curve During a Dosing Interval (AUCtau) of Esomeprazole After at Least 5 Days of Repeated Dose
Time Frame: 0, 0.5, 1, 1.5, 2, 3, 4 and 6 hours post-dose after at least 5 days of repeated dose
Population: All patients who had at least one plasma concentration data after administration of study drug without any protocol deviations that would have an impact on the pharmacokinetics (PK).
Measure: Mean (Standard Deviation); unit: μmol*h/L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 7 | 9 | 10 | 9 | 10
μmol*h/L | 7.04 (3.05) | 3.52 (2.35) | 11.05 (5.11) | 2.38 (1.74) | 5.82 (1.85)

18. Secondary Outcome: AUC From Time Zero to Time of Last Quantifiable Concentration (AUC0-t) of Esomeprazole After at Least 5 Days of Repeated Dose
Time Frame: 0, 0.5, 1, 1.5, 2, 3, 4 and 6 hours post-dose after at least 5 days of repeated dose
Population: All patients who had at least one plasma concentration data after administration of study drug without any protocol deviations that would have an impact on the PK.
Measure: Mean (Standard Deviation); unit: μmol*h/L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 9 | 10 | 10 | 9 | 10
μmol*h/L | 5.53 (3.69) | 3.09 (2.34) | 10.41 (4.55) | 1.99 (1.30) | 5.45 (1.78)

19. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Esomeprazole After at Least 5 Days of Repeated Dose
Time Frame: 0, 0.5, 1, 1.5, 2, 3, 4 and 6 hours post-dose after at least 5 days of repeated dose
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 9 | 10 | 10 | 9 | 10
μmol/L | 3.42 (2.09) | 2.09 (1.53) | 5.91 (2.19) | 1.09 (0.57) | 3.13 (1.36)

20. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Esomeprazole After at Least 5 Days of Repeated Dose
Time Frame: 0, 0.5, 1, 1.5, 2, 3, 4 and 6 hours post-dose after at least 5 days of repeated dose
Population: as for outcome 18
Measure: Median (Full Range); unit: hour
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 9 | 10 | 10 | 9 | 10
hour | 1.58 (2.09) [1.03 to 5.92] | 1.52 (1.53) [0.92 to 6.00] | 1.47 (2.19) [0.93 to 1.52] | 1.57 (0.57) [0.93 to 2.95] | 1.75 (1.36) [0.95 to 3.00]

21. Secondary Outcome: Elimination Half-life (t1/2) of Esomeprazole After at Least 5 Days of Repeated Dose
Time Frame: 0, 0.5, 1, 1.5, 2, 3, 4 and 6 hours post-dose after at least 5 days of repeated dose
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 7 | 9 | 10 | 9 | 10
hour | 0.80 (0.18) | 0.97 (0.55) | 1.08 (0.44) | 1.37 (0.88) | 1.06 (0.25)

22. Secondary Outcome: Apparent Total Clearance (CL/F) of Esomeprazole After at Least 5 Days of Repeated Dose
Time Frame: 0, 0.5, 1, 1.5, 2, 3, 4 and 6 hours post-dose after at least 5 days of repeated dose
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 7 | 9 | 10 | 9 | 10
L/h | 4.74 (1.92) | 12.44 (8.90) | 6.44 (3.37) | 23.33 (24.93) | 10.94 (3.64)

23. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Esomeprazole After at Least 5 Days of Repeated Dose
Time Frame: 0, 0.5, 1, 1.5, 2, 3, 4 and 6 hours post-dose after at least 5 days of repeated dose
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 7 | 9 | 10 | 9 | 10
L | 5.10 (1.24) | 16.56 (16.21) | 9.21 (4.00) | 44.73 (72.03) | 15.90 (4.42)

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the date of signing of informed consent to 8 weeks or withdrawal. Other adverse events were collected from the start of investigational drug administration to 8 weeks or withdrawal.
Description: During the administration period, the investigator/clinical research coordinator contacted the patient or patients' guardian (e.g. by phone) at least once in every week to confirm patient's health condition and compliance of study drug.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Serious Adverse Events (participants affected / at risk) | 2/10 | 0/10 | 0/10 | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 8/10 | 8/10 | 5/10 | 5/10 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=10) | Group 2 (N=10) | Group 3 (N=10) | Group 4 (N=10) | Group 5 (N=10)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=10) | Group 2 (N=10) | Group 3 (N=10) | Group 4 (N=10) | Group 5 (N=10)
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Mumps (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 4 | 2 | 1 | 3
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Varicella (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 2
Hordeolum (Eye disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs were prohibited to disclose all information related to this study without AstraZeneca approval before this study was completed.